CLINICAL TRIAL: NCT06739408
Title: Investigation of Protein Source and Its Impact on Response to Resistance Training
Brief Title: Protein Source and Resistance Training
Acronym: Pro-Train
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Elaine McCarthy, Principal Investigator, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ECM 3 (g) 22/10/2024
Record Dates: First submitted 2024-11-25; First posted 2024-12-18 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-12

CONDITIONS: Healthy; No Condition
Keywords: protein; skeletal muscle; resistance training; food; supplement; whey; meat
MeSH Terms: interventions — Whey Proteins; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lean Red Meat (Experimental): Cooked lean beef to provide approx 30g protein and isocalorically matched to be consumed 3x per week immediately following each resistance training session
  Interventions: Dietary Supplement: Lean red meat
- Whey Protein (Active Comparator): Whey protein to contain 30g of protein and isocalorically matched to be consumed 3x weekly immediately following each resistance training session
  Interventions: Dietary Supplement: Whey protein
- Maltodextrin (Placebo Comparator): Isocalorically matched but providing 0g protein to be consumed 3x per week immediately following each resistance training session
  Interventions: Dietary Supplement: Maltodextrin (Placebo)

INTERVENTIONS:
Dietary Supplement: Lean red meat — 30g of protein from lean beef.
  Arms: Lean Red Meat
Dietary Supplement: Whey protein — Whey protein to provide 30g protein
  Arms: Whey Protein
Dietary Supplement: Maltodextrin (Placebo) — Maltodextrin, to provide 0g protein but matched isocalorically
  Arms: Maltodextrin

SUMMARY:
The goal of this clinical trial is to investigate the role of whole food protein source compared with supplement forms in enhancing response to resistance exercise training in moderately active participants. The main question it aims to answer:

Whether wholefood protein (lean red meat) consumption is equivalent to supplementation in supporting muscle function and composition responses to resistance training? Whether wholefood protein consumption results in additional benefits to micronutrient status above that of supplementations? Researchers will compare both lean red meat and whey protein groups with an isocaloric maltodextrin control to see if protein intake enhanced response to resistance training.

* Participants will be randomized to consume one of three treatments: (1) lean red meat, (2) a whey protein supplement, or (3) an isocaloric maltodextrin control beverage following each resistance training session.
* Participants will complete a 12-week progressive resistance training programme consisting of 3 exercise sessions per week.
* Participants will undergo skeletal muscle performance testing by way of Vertical jump height, isokinetic strength tests and estimated one repetition maximum tests prior to and following the 12-week resistance training programme.
* Participants will undergo body composition assessment by way of bioelectrical impedance analysis, thigh muscle ultrasound and skinfold measurement prior to and following the 12-week resistance training programme.

DETAILED DESCRIPTION:
Background Protein supplements and particularly whey protein supplements are frequently consumed by athletes and recreationally active adults to achieve greater gains in muscle mass and strength as well as improved physical performance. Lean red meat has the equivalent essential amino acid and branched chain amino acids as whey protein, and additionally contains creatine, beta-alanine and several essential vitamins and minerals which are important for health and performance. Therefore, the preferential addition of lean red meat to the diet as opposed to whey protein supplements may provide the same and possibly greater benefits and would be in line with the recommended 'food first approach' endorsed by Sport Ireland and the World Anti-Doping Agency among others.

Aim The overall aim of this study is to explore whether lean red meat augments adaptation to resistance training in recreationally active young adults undergoing resistance training. Additionally, the investigators aim to investigate changes in nutritional intakes and status of selected micronutrients in response to increased consumption of lean red meat.

Methods

A total of n=72 recreationally active men and women (50% male) will be recruited to this single-blinded intervention study with a parallel design. Participants will be randomized to consume one of three treatments:

1. lean red meat,
2. a whey protein supplement, or
3. an isocaloric maltodextrin control beverage and will complete a 12-week resistance training programme.

Measurements: Body composition and muscle thickness will be measured using bioelectrical impedance analysis and ultrasound respectively. Additionally, skinfold measurements will be used to estimate body fat percentage. Vertical jump height, isokinetic strength and 1 repetition maximums will be completed to assess muscle contractile properties namely explosive and maximal strength. Blood pressure will also be measured at baseline and post intervention. Finally, dietary intake will be recorded at selected timepoints, and blood tests will be used to characterise status of selected micronutrients, blood lipids, and inflammation markers. All measures will be performed before and at the end of a 12-week resistance training intervention during which all participants will engage in resistance exercise 3 days per week and consume their assigned treatment on each of those training days.

Conclusion By investigating the impact of lean red meat on exercise adaptation and nutrition status of a number of selected micronutrients this study can contribute to the understanding of the role of lean red meat in performance nutrition. Additionally, this study can more broadly contribute to our understanding of the "food first" approach as it relates to recreationally active men and women.

ELIGIBILITY:
Inclusion Criteria:

* a. Aged between 18 to 35 years old. b. Have completed either no or low level only resistance training in the previous 6 months.

  c. Are not using any protein or performance/recovery enhancing supplements or willing to stop use for duration of the study.

  d. Willing to consume study treatment for duration of the study. e. Willing to perform resistance training. f. Must be able and willing to provide written informed consent to participate.

Exclusion Criteria:

1. Have any notable health concern or disability which may conceivably increase risk to the participant and/or affect outcomes.
2. Has performed resistance training in the past 6 months at a moderate or high level.
3. Is a smoker.
4. Is unwilling or unable to perform full body resistance training.
5. Is pregnant or planning to become pregnant during the study period.
6. Has a food allergy or intolerance that may place participant at risk to consume any of the study treatments.
7. Is post-menopausal or currently undergoing menopause.
8. Follows a vegetarian or meat-avoidant diet.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Isokinetic Dynamometry | 12-weeks from pre to post resistance training programme
  Change in primary leg Isokinetic lower limb strength will be measured using an isokinetic dynamometer (Biodex).

SECONDARY OUTCOMES:
Change to Fat Free Mass | 12-weeks from pre to post resistance training programme
  Bioelectric impedance analysis will be carried out to measure change from pre intervention to post intervention on fat free mass.
Thigh Muscle Ultrasound | 12-weeks from pre to post resistance training programme
  Ultrasound imaging will be carried out on the thigh muscles in the dominant leg before and after the intervention to determine changes in muscle thickness.
4-Site Skinfold Thickness | 12-weeks from pre to post resistance training programme
  4-site skinfold measurement will be assessed by an International Society for the Advancement of Kinanthropometry (ISAK) qualified anthropometrist to assess body composition changes.
Vertical Jump Height | 12-weeks from pre to post resistance training programme
  Vertical jump height will be recorded using the Leonardo mechanograph. The Leonardo mechanograph is a portable force plate system that records at a sampling rate of 800Hz and as such is a highly accurate method for recording jump height in a vertical jump.
Dietary Intake | 12-weeks from pre to post resistance training programme
  Dietary intake will be assessed using a 3-day food and drink diary. During both the baseline visit (week 0) and during the final week of the intervention (week 12), participants will be provided with a hard copy of the food and drink diary along with a digital weighing scale.
Change to LDL cholesterol | 12-weeks from pre to post resistance training programme
  A fasted venous blood sample will be taken by a suitably qualified and experienced nurse and assessed for changes in LDL cholesterol from pre intervention to post intervention
Change to serum ferritin status | 12-weeks from pre to post resistance training programme
  A fasted venous blood sample will be taken by a suitably qualified and experienced nurse. Participants will be asked to arrive to the human nutrition studies unit following an overnight fast on the morning of the baseline and endpoint visit. Participants will refrain from vigorous exercise for at least 24 hours prior to the blood draw. Blood sample will then be frozen for subsequent analysis of serum ferritin status
Change to total score on SAGIS questionnaire | 12-weeks from pre to post resistance training programme
  The change in total score obtained from the Structured Assessment of Gastrointestinal Symptoms (SAGIS) Questionnaire which is a validated tool used to assess gastrointestinal symptoms. Total symptom burden score can range from 0 to 88
Change to vitamin D status | 12-weeks from pre to post resistance training programme
  A fasted venous blood sample will be taken by a suitably qualified and experienced nurse. Participants will be asked to arrive to the human nutrition studies unit following an overnight fast on the morning of the baseline and endpoint visit. Participants will refrain from vigorous exercise for at least 24 hours prior to the blood draw. Blood sample will then be frozen for subsequent analysis of vitamin D status

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Studies Unit, University College Cork, Cork, Co. Cork, Ireland